CLINICAL TRIAL: NCT05632744
Title: Evaluation of CG-100 Intraluminal Bypass Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colospan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-113
Record Dates: First submitted 2022-11-08; First posted 2022-12-01 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CG-100 Intraluminal Bypass Device (Experimental): Subjects will be treated with CG-100 Intraluminal Bypass Device
  Interventions: Device: CG-100 Intraluminal Bypass Device

INTERVENTIONS:
Device: CG-100 Intraluminal Bypass Device — Subjects will be treated with the CG-100 Intraluminal Bypass Device

SUMMARY:
Evaluation of CG-100 Intraluminal Bypass device

ELIGIBILITY:
Inclusion Criteria (pre-operative):

1. Willing to comply with protocol-specified follow-up evaluations
2. 22-75 (inclusive) years of age at screening
3. Diagnosed with colorectal cancer
4. Has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Safety of the CG-100 Intraluminal Bypass Device | 10 days
  Assessment of Serious Adverse Events

SECONDARY OUTCOMES:
Safety of the CG-100 Intraluminal Bypass Device | 4 weeks
  Assessment of Serious Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No